CLINICAL TRIAL: NCT05252858
Title: A Pilot Study Investigating the nCAP Signal Relief Patch in Subjects Undergoing Primary Hip or Knee Replacement Surgery: A Prospective, Randomized, Open Label Trial
Brief Title: A Pilot Study Investigating the nCAP Signal Relief Patch in Subjects Undergoing Primary Hip or Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacques E. Chelly (Other)
Collaborators: nCap Medical (Industry)
Responsible Party: Sponsor-Investigator, Jacques E. Chelly, Professor of Anesthesiology and Perioperative Medicine and Orthopedic Surgery Director, Regional Anesthesiology Fellowship Program, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY22010018
Record Dates: First submitted 2022-02-03; First posted 2022-02-23 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Opioid Use; Pain, Post Operative
Keywords: Joint replacement surgery; Post operative pain management; Neuro capacitor
MeSH Terms: conditions — Pain, Postoperative | interventions — Standard of Care; Enhanced Recovery After Surgery

STUDY DESIGN:
Intervention Model Description: Single-center prospective, randomized, open label trial involving patients undergoing unilateral hip replacement and patients undergoing unilateral knee replacement that score <19 on the PROMIS Emotional Distress - Anxiety - Short Form 8a
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- nCAP + ERAS (Experimental): Participants will have the nCAP Signal Relief Patch and complete Enhanced Recovery After Surgery (ERAS) standard of care. After surgery, the subjects randomized to the intervention group will have the nCAP Signal Relief patch applied to their surgical dressing by a trained researcher in the immediate Post Anesthesia Care Unit (PACU).
  Interventions: Device: nCAP Signal Relief Patch; Other: Standard of Care
- ERAS alone (Active Comparator): Participants randomized into the control group will receive complete Enhanced Recovery After Surgery (ERAS) standard of care and no nCAP patch.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: nCAP Signal Relief Patch — nCAP Signal Relief Patch post-operatively applied to the subject's surgical dressing by a trained researcher in the immediate Post Anesthesia Care Unit (PACU)
  Other Names: nCAP; treatment patch
  Arms: nCAP + ERAS
Other: Standard of Care — Subjects will undergo surgery using the approved ERAS anesthetic and post-operative pain management protocols. At Shadyside Hospital, the ERAS Protocol for these subjects involves preoperative meloxicam 15mg PO, gabapentin 300mg PO, acetaminophen 1g PO. Intra-operative, patients receive a spinal block (bupivacaine) and propofol IV sedation. Postoperative pain medication is titrated to the individual patient's level of pain (0-10). 0.2 mg IV hydromorphone can be given for breakthrough pain, oxycodone 5mg PO for moderate pain (4-6) and oxycodone 10 mg PO for severe pain (7-10). Ketorolac 15 mg IV is given Q6H during the hospital stay. Discharge medication may be Norco 5-325mg as prescribed by the surgeon.
  Other Names: Enhanced Recovery After Surgery (ERAS)

SUMMARY:
Opioid addiction in post-operative patients is recognized but not fully understood; therefore, in order to address this growing crisis, it is essential to explore alternative approaches to managing pain and apply them to the surgical population. One potential non-opioid method of pain relief is the use of the nCAP Nano Patch, placed topically on the site of pain. The objective of this study is to investigate the efficacy of the nCAP Signal Relief Patch in reducing the perioperative opioid requirement in patients undergoing primary unilateral total hip or knee replacement surgery.

DETAILED DESCRIPTION:
After signing an informed consent, subjects will complete the PROMIS Emotional Distress - Anxiety - Short Form 8a before completing any other questionnaires. Subjects who have a raw score <19 will be enrolled in the study. Any subject who scores ≥ 19 will be considered a screen failure and excluded from the study.

Once the subject is enrolled, in the pre-operative holding area they will be asked to complete the Pain Catastrophizing Scale (PCS), the PROMIS® Emotional Distress-Depression - Short Form 8a, and the PROMIS® Item Bank v1.0 - Sleep- Disturbance - Short Form 8a prior to surgery. The subject will also conduct a baseline functionality test to assess mobility and strength in their leg. The functional recovery will be assessed by determining the patient ability to walk 100 feet, go up 5 steps and raise their leg on the day of surgery. Scores can be 0 (no ability to raise the leg), 1 (some ability to raise the leg), and 2 (complete ability to raise the leg). These assessments will take approximately 15 minutes to complete.

Once these assessments are completed, subjects will be equally randomized to the intervention group (nCAP Signal Relief Patch + standard of care) or control group (standard of care). Both the control group and intervention group will receive approved ERAS multimodal standard of care. Only the interventional group will receive an nCAP Signal Relief Patch. Randomization will occur by assigning the participant a subject ID number, and this ID number will correspond to a treatment allocation based on a pre-designed randomization schema.

Subjects will undergo surgery using the approved ERAS anesthetic and post-operative pain management protocols.

After surgery, the subjects randomized to the intervention group will have the nCAP Signal Relief patch applied to their surgical dressing by a trained researcher in the immediate Post Anesthesia Care Unit (PACU). Subjects will be made aware at the time of consent and throughout the trial that they can drop out of the study at any time if they do not like wearing the nCAP Signal Relief Patch. The control group will not receive a patch but will receive the standard of care ERAS protocol. Subjects in the intervention group will be instructed to keep the nCAP Signal Relief Patch on their surgical dressing to avoid the risk for skin irritation.

Pain using a Numerical Rating Scale (NRS) at rest and with movement as well as opioid requirement will be assessed in the PACU and daily until discharge.

Subjects assigned to the intervention group should keep the nCAP Signal Relief Patch in place for 72 hours on their surgical dressing and they will be instructed to remove it at home.

Once the subject is discharged, they will be contacted via email (REDCAP survey) on post-operative day 1, 2, 3, 7, 14, and 30 to record postoperative opioid consumption, non-opioid consumption, NRS pain at rest and with movement, pain catastrophizing (via Pain Catastrophizing Scale) sleep quality (via PROMIS Sleep Disturbance Short Form 8a) and to assess functional recovery. Functional recovery will be assessed by determining the patient ability to walk 100 feet, go up 5 steps and raise their leg on postoperative days 1, 2, 3, 7, 14, and 30 as well as the pain associated with it. Patient satisfaction with pain management after surgery will be assessed at the 30 day follow up (0- least satisfied to 10-most satisfied). Subjects who are contacted via REDCap to complete follow-up questionnaires and do not complete them on the day they are assigned will be contacted via telephone for a reminder. They will be considered lost to follow up after 3 phone attempts.

Information will be collected from the medical record, including: patient demographics, medical history, medication summary while in the hospital, as well as progress notes from the entire encounter to determine the existence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Scheduled for elective primary unilateral hip or knee replacement

Exclusion Criteria:

* Active clinical depression, anxiety or catastrophizing
* Raw score >19 on PROMIS Emotional Distress - Anxiety - Short Form 8a
* Active alcoholism (defined as daily use of more than 1 liter of wine and/or 3 or more shots of hard liquor) or drug abuse (defined as daily use of illicit drugs)
* Severe chronic pain condition that requires daily preoperative opioid dependence
* Total surgery revision, bilateral hip or nee replacement, other procedures under the same anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-10-08 (Actual); Study Completion 2022-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques E Chelly, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | nCAP + ERAS | ERAS Alone
Started | 38 | 31
Completed | 38 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | nCAP + ERAS | ERAS Alone | Total
Number analyzed (Participants) | 38 | 31 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 27 | 22 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (8.9) | 69.6 (9.0) | 68.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 30
  Male | 20 | 19 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 37 | 31 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 35 | 25 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 31 | 69
Weight [Mean (Standard Deviation); unit: kg] | 89.9 (10.6) | 89.1 (17.8) | 89.6 (14.2)
Height [Mean (Standard Deviation); unit: cm] | 170.0 (11.4) | 169.0 (11.5) | 169.5 (11.3)
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 31.4 (4.8) | 30.9 (4.7) | 31.2 (4.7)
Surgery Type [Count of Participants; unit: Participants]
  Total Knee Arthroplasty | 31 | 29 | 60
  Total Hip Arthroplasty | 7 | 2 | 9
PROMIS - Anxiety questionnaire [Mean (Standard Deviation); unit: T-score] — PROMIS (Patient-Reported Outcomes Measurement Information System) - Anxiety questionnaire raw scores were converted to T-score. PROMIS, measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For PROMIS measures, higher scores equals more of the concept being measured, for instance, higher anxiety. Thus a score of 60 is one standard deviation above the average referenced population. T-score of 60-70 is considered moderate levels of anxiety, and >70 is considered severe levels of anxiety.
  T-score | 48 (6.0) | 44.1 (7.5) | 46.2 (7.0)
PROMIS - Emotional Distress - Depression questionnaire [Mean (Standard Deviation); unit: T-score] — Measure Description: PROMIS (Patient-Reported Outcomes Measurement Information System) - Emotional Distress - Depression questionnaire raw scores were converted to T-score. PROMIS, measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. Higher scores equals more of the concept being measured, for instance, higher depression. Thus a score of 60 is one standard deviation above the average referenced population. T-score of 60-70 is considered moderate, and >70 is considered severe levels of depression.
  T-score | 41.9 (7.1) | 40.4 (4.7) | 41.3 (6.2)
PROMIS - Sleep Disturbance questionnaire [Mean (Standard Deviation); unit: T-score] — Measure Description: PROMIS (Patient-Reported Outcomes Measurement Information System) - Sleep Disturbance questionnaire raw scores were converted to T-score. PROMIS, measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. Higher scores equals more of the concept being measured, for instance, higher levels of sleep disturbance. Thus a score of 60 is one standard deviation above the average referenced population.
  T-score | 51.4 (7.0) | 47.4 (9.3) | 49.6 (8.3)
Pain Catastrophizing scale [Mean (Standard Deviation); unit: units on a scale] — Pre-operative pain ratings will be measured by the assessment of the participant's answers to the Pain Catastrophizing Scale questionnaire. There are 14 statements related to pain that participants will record experiencing on a scale of 0 being experienced not at all to 4 being experienced all of the time. The lowest possible score is 0 and the highest possible score is 56. Higher scores present a worse outcome.
  units on a scale | 5.8 (6.1) | 6.8 (8.4) | 6.3 (7.2)
Functional Recovery Test [Mean (Standard Deviation); unit: units on a scale] — Patients completed the Functional Recovery Test questionnaire to evaluate their ability to walk, climb stairs, and perform leg raises. Scores ranged from 0-4, with higher scores indicating better functional status.
  units on a scale | 3.7 (0.6) | 3.5 (1.0) | 3.6 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of the nCAP Signal Relief Patch in Affecting Perioperative Opioid Requirement
Description: The primary endpoint will be to prospectively investigate the efficacy of the nCAP Signal Relief Patch in reducing perioperative opioid requirement in opioid-naïve patients undergoing primary unilateral total hip or knee replacement surgery using currently SHY ERAS anesthesia protocol. This is reported in consumption of oral morphine mg equivalents (OME) from the day of surgery up to day 30 post-operative. Opioid requirement will be estimated following the placement of the patch.
Time Frame: Day of surgery up to 30 days post-operative
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | nCAP + ERAS | ERAS Alone
Number analyzed (Participants) | 38 | 31
MME | 82.1 (80.3) | 102.6 (74.0)

2. Secondary Outcome: Pre-operative Emotional Distress Related to Anxiety
Description: Pre-operative emotional distress related to anxiety will be measured by assessment of participant's answers to the PROMIS Emotional Distress -Anxiety- Short Form 8a questionnaire prior to surgery. There are 8 questions about how the participants may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher T-scores present a worse outcome for anxiety. For the adult PROMIS Anxiety 8a short form values reported, the participants raw scores are converted to T-scores and then averaged.
Time Frame: Screening visit
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | nCAP + ERAS | ERAS Alone
Number analyzed (Participants) | 38 | 31
T-score | 48.0 (6.0) | 44.1 (7.5)

3. Secondary Outcome: Post-operative Change in Emotional Distress Related to Anxiety
Description: Post-operative emotional distress related to anxiety will be measured by assessment of participant's answers to the PROMIS Emotional Distress -Anxiety- Short Form 8a questionnaire. There are 8 questions about how the participants may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher T-scores present a worse outcome for anxiety. For the adult PROMIS Anxiety 8a short form values reported, the participants raw scores are converted to T-scores and then averaged.
Time Frame: Day of surgery up to 30 days post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | nCAP + ERAS | ERAS Alone
Number analyzed (Participants) | 38 | 31
units on a scale | 9.85 (3.31) | 9.68 (2.93)

4. Secondary Outcome: Pre-operative Emotional Distress Related to Depression
Description: Pre-operative emotional distress related to depression will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Depression-Short Form questionnaire prior to surgery. There are 8 questions about how the participant may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher T-scores present a worse outcome for depression. For the adult PROMIS Depression 8a short form values reported, the participants raw scores are converted to T-scores and then averaged.
Time Frame: Screening visit
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | nCAP + ERAS | ERAS Alone
Number analyzed (Participants) | 38 | 31
T-score | 41.9 (7.1) | 40.4 (4.7)

5. Secondary Outcome: Post-operative Change in Emotional Distress Related to Depression
Description: Post-operative emotional distress related to depression will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Depression-Short Form questionnaire. There are 8 questions about how the participant may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher T-scores present a worse outcome for depression. For the adult PROMIS Depression 7a short form values reported, the participants raw scores are converted to T-scores and then averaged.
Time Frame: Day of surgery up to 30 days post-operative
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | nCAP + ERAS | ERAS Alone
Number analyzed (Participants) | 38 | 31
T-score | 42.25 (6.78) | 41.78 (6.48)

6. Secondary Outcome: Pre-operative Sleep Disturbance
Description: Pre-operative sleep disturbance will be measured by assessment of the participant's answers to the PROMIS item Bank v1.0 - Sleep Disturbance - Short Form 8a. There are 8 questions about how the participant may have felt about their sleep quality in the past 7 days. The scale for 1 question is very poor in the past 7 days to very good in the past 7 days. Higher T-scores present a worse outcome for sleep disturbance. For the adult PROMIS Sleep Disturbance 8a short form values reported, the participants raw scores are converted to T-scores and then averaged.
Time Frame: Screening visit
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | nCAP + ERAS | ERAS Alone
Number analyzed (Participants) | 38 | 31
T-score | 51.4 (7.0) | 47.4 (9.3)

7. Secondary Outcome: Post-operative Change in Sleep Disturbance
Description: Post-operative sleep disturbance will be measured by assessment of the participant's answers to the PROMIS item Bank v1.0 - Sleep Disturbance - Short Form 8a. There are 8 questions about how the participant may have felt about their sleep quality in the past 7 days. The scale for 1 question is very poor in the past 7 days to very good in the past 7 days. Higher T-scores present a worse outcome for sleep disturbance. For the adult PROMIS Sleep Disturbance 8a short form values reported, the participants raw scores are converted to T-scores and then averaged.
Time Frame: Day of surgery up to 30 days post-operative
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | nCAP + ERAS | ERAS Alone
Number analyzed (Participants) | 38 | 31
T-score | 49.86 (8.81) | 49.11 (9.12)

8. Secondary Outcome: Average Score of Functionality at Baseline
Description: Functionality at baseline is assessed by asking the patient the following 3 questions:
  1. Are you able to walk 100 feet (No=0, or Yes = 1),
  2. Are you able to move up to five steps (No=0, or Yes = 1), and
  3. Are you able to raise your leg (No = 0, some = 1, completely = 2).
  The total score could vary from 0 to 4. Higher scores indicate better functional status.
Time Frame: Screening visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | nCAP + ERAS | ERAS Alone
Number analyzed (Participants) | 38 | 31
units on a scale | 3.7 (0.6) | 3.5 (1.0)

9. Secondary Outcome: Average Score of Functionality Post-Operative
Description: Functionality post-operative is assessed by asking the patient the following 3 questions:
  1. Are you able to walk 100 feet (No=0, or Yes = 1),
  2. Are you able to move up to five steps (No=0, or Yes = 1), and
  3. Are you able to raise your leg (No = 0, some = 1, completely = 2).
  The total score could vary from 0 to 4.
Time Frame: Day of surgery up to 30 days post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | nCAP + ERAS | ERAS Alone
Number analyzed (Participants) | 38 | 31
units on a scale | 2.8 (0.2) | 2.7 (0.1)

10. Secondary Outcome: Pre-operative Pain Rating Using the Pain Catastrophizing Scale
Description: Pre-operative pain ratings will be measured by the assessment of the participant's answers to the Pain Catastrophizing Scale questionnaire. There are 14 statements related to pain that participants will record experiencing on a scale of 0 being experienced not at all to 4 being experienced all of the time. The lowest possible score is 0 and the highest possible score is 56. Higher scores present a worse outcome.
Time Frame: Screening visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | nCAP + ERAS | ERAS Alone
Number analyzed (Participants) | 38 | 31
units on a scale | 5.8 (6.1) | 6.8 (8.4)

11. Secondary Outcome: Change in Post-operative Pain Rating Using the Pain Catastrophizing Scale
Description: Post-operative pain ratings will be measured by the assessment of the participant's answers to the Pain Catastrophizing Scale questionnaire. There are 14 statements related to pain that participants will record experiencing on a scale of 0 being experienced not at all to 4 being experienced all of the time. The lowest possible score is 0 and the highest possible score is 56. Higher scores present a worse outcome
Time Frame: Day of surgery up to 30 days post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | nCAP + ERAS | ERAS Alone
Number analyzed (Participants) | 38 | 31
units on a scale | 4.3 (5.8) | 4.6 (6.3)

12. Secondary Outcome: Length of Hospital Stay
Description: Evaluate time to hospital discharge from out of OR time. This outcome measure will be measured via averaged hours to hospital discharge.
Time Frame: Day of surgery up to 30 days post-operative
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | nCAP + ERAS | ERAS Alone
Number analyzed (Participants) | 38 | 31
hours | 31.72 (22.0) | 40.85 (36.23)

13. Secondary Outcome: Change in Post-operative Pain Using a Numerical Rating Scale
Description: Numerical Rating Scale (NRS) Pain scores on a scale from 0-10, with 0 being no pain, 5 being moderate pain and 10 being the worst imaginable pain. The outcome measure is an area under the curve from POD 1 to POD 30, with the unit of pain per day being measure 0-300 (scale of 0-10 for 30 days).
Time Frame: Days 1-30 post-operative
Measure: Mean (Standard Deviation); unit: Scores X Day
Arm/Group | nCAP + ERAS | ERAS Alone
Number analyzed (Participants) | 38 | 31
Scores X Day | 59.4 (41.6) | 101.5 (75.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of enrollment to POD 30 (end of study)
Arm/Group | nCAP + ERAS | ERAS Alone
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/31
Other Adverse Events (participants affected / at risk) | 0/38 | 0/31

LIMITATIONS AND CAVEATS:
Although the present study is the first prospective, randomized study on the use of the NeuroCupleTM device, our data will need to be confirmed by a larger randomized placebo-controlled study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT05252858/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT05252858/SAP_003.pdf
  • Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT05252858/ICF_002.pdf